CLINICAL TRIAL: NCT02039518
Title: Randomized Controlled Trial of Gemcitabine Maintenance Treatment in Patients With Extensive SCLC Patients Receiving Etoposide Combined With Platinum Based First-line Chemotherapy
Brief Title: Study of Gemcitabine Maintenance Treatment in Patients With Extensive SCLC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xianghua Wu, Associate Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WXH-gemcitabine-SCLC
Record Dates: First submitted 2013-12-30; First posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Small Cell Lung Cancer
Keywords: Progression free Survival
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemcitabine (Experimental): gemcitabine 1000mg/m2，d1，d8，Q3W
  Interventions: Drug: gemcitabine
- observation group (Other): observation
  Interventions: Other: observation group

INTERVENTIONS:
Drug: gemcitabine — gemcitabine 1000mg/m2，d1，d8，Q3W
  Other Names: gemcitabine 1000mg/m2，d1，d8，Q3W
  Arms: gemcitabine
Other: observation group — observation group
  Arms: observation group

SUMMARY:
The purpose of this study is to Evaluate and compare safety and efficacy of Gemcitabine Maintenance Treatment in Patients With Extensive SCLC Patients Receiving Etoposide Combined With Platinum Based First-line Chemotherapy

DETAILED DESCRIPTION:
from the first cycle of treatment (day one) to two month after the last cycle

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. PS=0,1,2
3. Patients who were diagnosed by the histologic, cytologic diagnosis of extensive small cell lung cancer
4. Patients received Etoposide combined with platinum based first-line chemotherapy 6 cycles and there is evidence show the patent is PR/CR/SD
5. Expected lifetime>12 weeks
6. Signed written informed consent

Exclusion Criteria:

Small cell lung cancer non small cell hybrid Women during pregnancy or lactation previously treated with two or more than two kinds of treatment Any non remission of >CTCAE caused tumor treatment past grade 2 toxicity Ccr<30 ml/min (calculated by Cockcroft-Gault formula) hepatic insufficiency：

1. Tbil> 1.5×ULN
2. ALT and AST > 2.5×ULN (Patients with liver metastasis>5×ULN) Alkaline phosphatase>2.5 ×ULN(Patients with liver metastasis>5×ULN)
3. Severe symptomatic heart disease
4. Symptomatic brain metastases
5. In the last 5 years have been or are suffering from other histological types of malignant tumor
6. There are serious or uncontrolled systemic diseases
7. During the study period planned radiotherapy on target lesion
8. During the study period, plans to use other antineoplastic therapy
9. Clinical study on treatment of 30 days beginning period prior to participate in any study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Overall Officials: WU X HUA, DOCTOR, Principal Investigator — Fudan University
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China